CLINICAL TRIAL: NCT03419169
Title: Light Load Blood Flow Restriction Versus Heavy Load Resistance Training in the Post-operative Rehabilitation of Anterior Cruciate Ligament Reconstruction Patients
Brief Title: Light Load Blood Flow Restriction Training in Anterior Cruciate Ligament Reconstruction Patient Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: St. Mary's University, Twickenham (Other)
Responsible Party: Principal Investigator, Luke Hughes, Principal Investigator, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/YH/0066
Record Dates: First submitted 2018-01-18; First posted 2018-02-01 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Patient; Rehabilitation; Ligament reconstruction; Surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to one of two groups: 1) Light load BFR resistance training; or 2) Heavy load resistance training. An independent member of the research team will carry out block randomisation using opaque envelopes containing slips of paper. Each envelope will contain four slips (Two x BFR group and two x heavy load group), thus patients will be randomised in groups of four.
Who Masked: Outcomes Assessor
Masking Description: The assessor of all outcome measures will be masked as to which group patients have been assigned. Patient information will be coded using a numerical system by and independent member of the research team during the course of the study and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Light load BFR resistance training (Experimental): This arm of the clinical trial will involve eight weeks of twice weekly light load resistance training with BFR. Patients in this arm will complete four sets (30, 15, 15 and 15 repetitions, respectively) of unilateral leg press exercise at 30% of predicted one repetition maximum. BFR will be applied at 80% of total limb arterial occlusive pressure. Both legs will be trained, with the affected limb trained first and the unaffected limb matched for volume at a relative percentage of one repetition maximum. Both legs will be trained with BFR.
  Interventions: Device: Light load BFR resistance training
- Heavy load resistance training (Active Comparator): This arm of the clinical trial will involve eight weeks of twice weekly heavy load resistance training. Patients in this arm will complete three sets of ten repetitions of unilateral leg press exercise at 70% of predicted one repetition maximum. Both legs will be trained, with the affected limb trained first and the unaffected limb matched for volume at a relative percentage of one repetition maximum.
  Interventions: Procedure: Heavy load resistance training

INTERVENTIONS:
Device: Light load BFR resistance training — A novel training light load resistance training modality.
  Arms: Light load BFR resistance training
Procedure: Heavy load resistance training — A common form of resistance training used for rehabilitation within the National Health Service.
  Arms: Heavy load resistance training

SUMMARY:
This study is examining the post-operative rehabilitation of anterior cruciate ligament (ACL) reconstruction patients within the National Health Service (NHS). It will compare the effectiveness of two resistance training protocols, light load blood flow restriction (BFR) training and heavy load training, on improving multiple aspects important to the rehabilitation process in this patient demographic, whilst also examining the feasibility of this novel training modality. It is hypothesised that light load BFR training will be equally effective as heavy load training, but more tolerable for patients.

DETAILED DESCRIPTION:
Light load BFR training is an effective rehabilitation tool for improving strength in individuals suffering clinical muscle weakness (Hughes et al. 2017). This is a single blinded, randomised controlled clinical trial, comprised of a two (group) by five (time) between-subjects repeated measures design. This study will place within the NHS at University College London Hospital (UCLH). Eligible patients from the orthopaedic department theatre lists of four orthopaedic surgeons at UCLH will be contacted prior to surgery via phone call and sent the patient information sheet and schematic outlining the study. Patient clinical history and documentation will be screened initially by the principle researcher followed by screening over the phone upon contact. Patients who are willing to participate will then be invited to the hospital for a full health screening appointment following provision of written informed consent, in compliance with the Declaration of Helsinki, 7th version, October 2013.

Baseline assessment of all outcome measures will take place at the pre-surgery screening appointment. Patient will then undergo their surgery. Following two weeks of recovery, repeat assessment of outcome measures will take place once patients achieve the following criteria for beginning strength rehabilitation, as developed by Cavanaugh and Powers (2017): 1) Able to unilaterally weight bear without pain; 2) Able to perform a single leg raise without quadriceps lag; 3) Have a range of motion (ROM) of 0-90 degrees; and 4) Have minimal swelling. Patients will then be allocated to one f the two training intervention groups and undergo eight weeks of twice weekly unilateral leg press training. Training sessions include five minutes of light cycling at a free cadence on a stationary ergometer for both groups, followed by the respective leg press protocols. Repeat assessment of outcome measures will take place mid-training (between weeks four and five) and post-training. Ratings of perceived pain and exertion, blood pressure and any adverse events will be recorded at all training and assessment sessions. All outcomes will also be assessed at 3 and 6 month follow up assessments. Pain will also be assessed 24 hours after every training session. During the study, all participants will see their assigned physiotherapist fortnightly (as per standard hospital protocol) and receive individualised programmes focussing on improving ROM, balance and minimising swelling.

BFR will be achieved using the Delfi Easy-fit variable contour tourniquet cuff (11.5 cm x 86 cm x 5 mm) connected to the automatic personalised tourniquet system (PTS) device (Delfi Medical, Vancouver, British Columbia, Canada). The Delfi PTS for BFR is equipped with the capability of automatically measuring limb occlusive pressure (LOP) and calculating the personalised tourniquet pressure, comprised of a dual-purpose personalised tourniquet cuff and a personalised tourniquet instrument containing LOP calculation sensors and software. The PTS system connected to the tourniquet cuff increases the cuff pressure in stepwise increments, analyses the pneumatic pressure pulsations in the cuff bladder by the arterial pressure pulsations at each cuff pressure increment, and uses these characteristics to determine LOP.

The primary outcome measure of muscle strength was used for calculating the required sample size. Based on previous data regarding muscle strength increases in light load BFR resistance training studies in clinical populations, to achieve a power of 80% at an alpha level 0.05, a total of 28 participants is required to detect a meaningful effect. Based on hospital record of rehabilitation programmes, a drop-out rate of 10% can be expected during the course of rehabilitation programmes. Therefore, a total of 30 participants will be recruited.

All data will be stored on the NHS password protected server at UCLH as per hospital and NHS ethical requirements. Data from drop-outs will not be included in the final analysis. Descriptive statistics (mean ± standard deviation) will be used to summarise adherence rates, exercise session attendance, training volume any adverse events. All statistical analysis will be performed with IBM Statistical Package for the Social Sciences (SPSS) Version 22.0 (IBM Corp, Chicago Illinois, United States of America). All data will be presented as means ± standard deviation with 95% confidence intervals unless stated otherwise. Normal distribution of data will be assessed using Shapiro-Wilks test (p>0.05). Ten repetition maximum strength, muscle size measures, self-reported physical function measures and functional performance will each be analysed using 2 x 5 (rehabilitation intervention x TP) repeated measures analysis of variance (ANOVA)s. Isokinetic strength and knee ligament laxity will be assessed using 2 x 3 (rehabilitation intervention x TP) repeated measures ANOVAs. Perceptual responses for ratings of perceived exertion and pain will be assessed using 2 x 16 (rehabilitation intervention x exercise session) repeated measures ANOVAs. For any statistically significant two-way interaction, one-way repeated measures ANOVAs with Bonferroni correction will be used to examine simple main effects. Non-normally distributed data will be analysed using the non-parametric Friedman test. Alpha significance will be set a priori p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Registered patient of University College London Hospitals
2. Over 18 years of age
3. Present with a unilateral ACL tear

5. Scheduled for reconstructive surgery 6. Have the mental capacity to make informed decisions

Exclusion Criteria:

1. Multiple ligamentous ruptures or trauma
2. Rheumatoid arthritis or significant comorbidities
3. Presence or history of cardiovascular, pulmonary, respiratory of neurological disease
4. Intraarticular injections into the knee in the preceding 6 months
5. History of deep vein thrombosis or vascular pathology in any lower limb
6. Current use of anticoagulant medications or other medications that may affect blood flow or fluid exchange
7. Hypertension (>140/80 mmHg)
8. Inability to follow instructions for rehabilitation classes (e.g. advanced dementia)
9. Scheduling for post-operative leg bracing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in ten repetition maximum strength | Throughout study completion, up to one year
  Unilateral isotonic muscle strength, measured in kilograms.
Change in isokinetic strength | Throughout study completion, up to one year
  Unilateral peak torque at 60°/second, 150°/second, and 300°/second, measured in newton-metres.

SECONDARY OUTCOMES:
Muscle thickness, measured in centimetres | Throughout study completion, up to one year
  Thickness of the vastus lateralis muscle
Pennation angle of muscle fibres, measured in degrees (°) | Throughout study completion, up to one year
  Angle of fibres in the vastus lateralis muscle
Fascicle length, measured in centimetres | Throughout study completion, up to one year
  Length of fascicles in the vastus lateralis muscle
International Knee Documentation Committee subjective knee form | Throughout study completion, up to one year
  Used to assess symptoms and function in daily living activities
Knee Injury and Osteoarthritis Outcome Score | Throughout study completion, up to one year
  Used to assess participant's opinion of their knee and associated problems
Lower Extremity Functional Scale to assess performance in functional tasks | Throughout study completion, up to one year
  Used to assess patient's ability to perform everyday tasks, including walking and stair climbing. It contains 20 questions each with a scoring scale of 0-4 and a test-retest reliability of 0.88 to 0.94. The scores of each question will be summed to get a total score out of 80, with lower scores indicating greater functional disability. The minimal detectable change will be set at 9 scale points.
Lysholm knee scoring scale to assess performance in functional tasks. | Throughout study completion, up to one year
  Used to evaluate outcomes of the surgery. It comprises 8 items, including: limp, support, locking, instability, pain, swelling, stair climbing and squatting. Each item is scored differently - scores will be summed to give a total out of 0-100 (where 100 indicates no symptoms or disability) and categorised as excellent (95-100), good (84-94), fair (65-83), and poor (≤64).
Tegner activity scale for grading patient activity level | Throughout study completion, up to one year
  Used to grade participant activity level. The scale ranges from 0-10, with 0 representing sick leave or disability pension because of knee problems, and 10 corresponding to participation in national and international elite competitive sports. Minimum clinically importance difference will be set at 1.
Physical functional performance | Throughout study completion, up to one year
  Star-excursion balance test of dynamic knee joint stability, measured in centimetres
Knee ligament laxity | Throughout study completion, up to one year
  Laxity of the knee, measured in pounds.
Borg's (1998) rating of perceived pain scale for assessing pain during exercise. | During all testing sessions, between sets during all training sessions over the eight week training period, and 24 hours post-training for every training session.
  Used to measured the patient's perceived pain during exercise. The scale ranges from 0 to 10. Patients will be informed that a rating of 0 means they felt no pain, and 10 is their reference point which represents their previous worst felt pain/discomfort, and that they can give a score of 11 if the pain is worse than any they have ever felt before.
Borg's (1998) rating of perceived exertion scale for assessing exertion during exercise. | During all testing sessions and between sets during all training sessions over the eight week training period.
  Used to measured the patient's perceived exertion during exercise. The scale ranges from 6-20. It will be explained to patients that a rating of 6 meant they felt no exertion, and 20 meant they were giving maximal effort and could not exert themselves any further.
Blood pressure | Pre-exercise and 5 minutes post-exercise for all training sessions over the eight week training period
  Systolic and diastolic blood pressure, measured in millimetres of mercury using an automatic device.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Patterson, PhD, Principal Investigator — St. Mary's University, Twickenham; Fares Haddad, Principal Investigator — University College London Hospital
Locations (2):
- United Kingdom (2):
  - University College London Hospitals, London
  - St. Mary's University, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Cavanaugh JT, Powers M. ACL Rehabilitation Progression: Where Are We Now? Curr Rev Musculoskelet Med. 2017 Sep;10(3):289-296. doi: 10.1007/s12178-017-9426-3. PMID 28791612
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714